CLINICAL TRIAL: NCT02086149
Title: Aerobic Exercise for Smokers With Depressive Symptomatology
Brief Title: Exercise for Depressed Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1304-001; R01CA173551 (NIH)
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Tobacco Smoking; Smoking Cessation
Keywords: Quit smoking; Exercise; Tobacco; Smoking
MeSH Terms: conditions — Tobacco Smoking; Smoking Cessation; Motor Activity; Smoking | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): 12-week moderate-intensity behavioral exercise intervention (AE)
  Interventions: Behavioral: Aerobic Exercise
- Health Education (Active Comparator): 12-week health education control
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Aerobic Exercise — 12-week moderate-intensity behavioral exercise intervention. Weekly sessions with an exercise physiologist who will also assign weekly exercise goals. Two month course of the nicotine patch initiated during week 5.
  Arms: Exercise
Behavioral: Health Education — 12-week health education control. Weekly sessions about 12 different topics related to the health effects of smoking, led by an expert in smoking cessation.
  Arms: Health Education

SUMMARY:
The purpose of this study is to test the effect of a moderate-intensity aerobic exercise intervention for helping individuals with elevated depressive symptoms to quit smoking. The investigators expect that this project will contribute much needed knowledge about the role that aerobic exercise can play in smoking cessation. The long-term goal of this program of research is to disseminate an effective, aerobic exercise (AE) intervention for smoking cessation that can be readily adopted by smokers with elevated depressive symptoms, including those with current major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

1. are between 18 and 65 years of age
2. are current smokers (i.e., smoking at least 10 cigarettes per day)
3. have currently elevated depressive symptoms (CES-D ≥ 6)
4. are sedentary, i.e., have not participated regularly in aerobic exercise (for at least 90 minutes per week during the past three months)

Exclusion Criteria:

1. DSM-IV diagnosis of current mania
2. DSM-IV diagnosis of bipolar rapid cycling
3. lifetime history of psychotic disorder or DSM-IV diagnosis of current psychotic symptoms
4. DSM-IV diagnosis of current substance abuse or dependence in the past 6 months
5. DSM-IV diagnosis of anorexia or bulimia nervosa
6. current suicidality or homicidality
7. marked organic impairment
8. current use of antidepressant medication for less than 3 months or change in antidepressant medication or dosage in the past 3 months,
9. physical disabilities or medical problems that would prevent or hinder participation in a program of moderate intensity exercise (i.e., physician denied medical clearance)
10. current pregnancy or intent to become pregnant during the next 12 weeks
11. contraindications for use of the nicotine patch (e.g., pregnancy, recent myocardial infarction, arrhythmia, angina, untreated hypertension, untreated diabetes, and previous adverse reaction to the patch)
12. current illness or medications that may alter proposed inflammatory markers (e.g., acute infection, immune disorders, aspirin)
13. current use of any pharmacotherapy or other treatment for smoking cessation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation | 1 year
  Abstinence from smoking verified biochemically (saliva cotinine)

CONTACTS AND LOCATIONS:
Overall Officials: Ana M. Abrantes, Ph.D., Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States